CLINICAL TRIAL: NCT03634579
Title: Magnetic Resonance Imaging (MRI) Guided Focal Laser Interstitial Thermal Ablation of Localized Prostate Cancer
Brief Title: MRI Guided Prostate Cancer Focal Laser Ablation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding for continuation.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Sherif G. Nour, Associate Professor of Radiology, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00094958
Record Dates: First submitted 2018-07-19; First posted 2018-08-16 (Actual); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: Cancer/Carcinogenesis; Laser Treatment; Magnetic Resonance Imaging (MRI); Radiology
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Carcinogenesis

STUDY DESIGN:
Intervention Model Description: Prospective, Interventional, Single-Arm, Unblinded trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- MRI-guided focal laser ablation (Experimental): Subjects will undergo MRI Guided Focal Laser Interstitial Thermal Ablation of localized low and intermediate risk prostate cancer.
  Interventions: Device: MRI Guided Focal Laser Interstitial Thermal Ablation

INTERVENTIONS:
Device: MRI Guided Focal Laser Interstitial Thermal Ablation — The procedure is done under general anesthesia. Laser fiber placement will be performed by one of two approaches (Trans gluteal or trans rectal) based on the target location within the prostate gland. When the needle position is deemed satisfactory, a 1.5-cm-active tip diode laser fiber will be introduced within an internally cooled catheter through the introducing sheath.
  The catheter tip location will be confirmed on Turbo Spin-Echo (TSE) T2-weighted images in the axial and sagittal oblique planes.The introducer sheath will be withdrawn to allow contact of the active laser tip with the lesion. A laser test dose will be done at 9 Watts for about 30 seconds to confirm the site of fiber placement with the subsequent delivery of full dose ablation at 12-27 Watts. Ablation duration is determined based on real time feedback of response using real time temperature and damage estimate maps.

SUMMARY:
The study is a prospective, single-arm, non-randomized, unblinded trial to determine the safety and efficacy of MRI guided focal laser ablation of localized low and intermediate risk prostate cancer. All subjects meeting the inclusion exclusion criteria and are enrolled will undergo a MRI guided focal laser ablation procedure. The primary aim of the study is to study the safety and efficacy of the procedure.

DETAILED DESCRIPTION:
Prostate cancer should be viewed as a spectrum of diseases ranging from a very indolent low-risk process to an aggressive high-risk potentially fatal disease. Active surveillance has been introduced as an alternative treatment to patients with low- risk prostate cancers.Focal therapy techniques have been introduced in prostate cancer to destroy the tumor itself with adequate safety margin with the advantage of preserving the surrounding non-cancerous tissue. Thus maintaining disease control at acceptable levels, while minimizing complications.

With the advent of multiparametric MRI (Mp-MRI), it is now possible to identify suspicious prostate gland focal lesions, determining their extent and targeting them for biopsy and focal ablation. Laser interstitial thermal therapy (LITT) is well suited for MRI environment. Laser fibers are flexible so they can fit into the MRI gantry. Laser has been shown to produce homogenous tissue necrosis that can be monitored by real time temperature maps, a feature that facilitates effective and safe ablation.

20 subjects with localized low and intermediate risk prostate cancer that meet the inclusion and exclusion criteria will be enrolled. During baseline evaluation, subjects will undergo lab tests, MR imaging, and will complete QOL questionnaires. Subsequently, subjects will undergo the Magnetic Resonance Imaging (MRI) Guided Focal Laser Interstitial Thermal Ablation procedure. Subjects will be followed immediately after the procedure, at 3 weeks, 3 months, 6 months, one year and two years after procedure for adverse events and recurrence of prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with primary organ confined prostate cancer (≤T2c) and Gleason score ≤4+3=7

  * Lesions visible on multiparametric MRI and subsequently diagnosed by targeted MRI guided biopsy

Exclusion Criteria:

* Multifocal intra-prostatic disease, defined as the presence the presence of ≥ 3 non- contiguous pathologically proven foci of cancer.
* Gleason score >4+3=7.
* Extracapsular spread.
* Nodal or distant metastasis
* Contraindications to MRI or general anesthesia.
* Uncorrectable Coagulopathy.
* Refusal of participation.
* Lesions not visualized on the multiparametric MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif G Nour, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRI-guided Focal Laser Ablation
Started | 9
Completed | 0
Not Completed | 9
Not completed — study termination | 9

BASELINE CHARACTERISTICS:
Arm/Group | MRI-guided Focal Laser Ablation
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Recurrences of Prostate Cancer at the End of 1 Year Among the Subjects Treated With MRI Guided Focal Laser Interstitial Thermal Ablation
Description: Efficacy is assessed by recurrence rate at 1 year, defined as the number of recurrences divided by the number of patients treated with MRI Guided Focal Laser Interstitial Thermal Ablation
Time Frame: Up to 12 months
Population: Data were not collected/analyzed due to the study termination
Arm/Group | MRI-guided Focal Laser Ablation
Number analyzed (Participants) | 0

2. Primary Outcome: Percentage of Grade 3 or Higher Complications as Defined as National Cancer Institute's Common Toxicity Criteria Version 4 Among the Subjects Treated With MRI Guided Focal Laser Interstitial Thermal Ablation
Description: Safety is assessed by percentage of grade 3 or higher complications or adverse events (AE) as defined as National cancer institute's common toxicity criteria version 4: incontinence or urinary retention necessitating surgical intervention or new-onset erectile dysfunction not responsive to medication.Grade refers to the severity of the AE. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.Grade 2 Moderate; minimal, local or non invasive intervention indicated; limiting age appropriate instrumental ADL. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: Up to 24 months
Measure: Number; unit: percentage of grade 3 or higher complica
Arm/Group | MRI-guided Focal Laser Ablation
Number analyzed (Participants) | 9
percentage of grade 3 or higher complica | 0

3. Primary Outcome: Number of Subjects Experienced Change in Erectile Function
Description: Change in erectile function is assessed using Sexual Health Inventory For Men (SHIM) for erectile function. There are 5 questions and each question has 5 possible responses. If the patient's score is 21 or less, erectile dysfunction (ED) is present.
Time Frame: 3 weeks follow up
Measure: Count of Participants; unit: Participants
Arm/Group | MRI-guided Focal Laser Ablation
Number analyzed (Participants) | 9
Participants | 1

4. Primary Outcome: Number of Subjects Experienced Change in Urinary Function
Description: Urinary function will be assessed using International Prostate Symptom Score (IPSS) assessment for urinary function. The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions (maximum score 35) concerning urinary symptoms and one question concerning quality of life. Any score > 1 indicates presence of urinary dysfunction, higher score indicates increased severity.
Time Frame: 3 weeks follow up
Measure: Count of Participants; unit: Participants
Arm/Group | MRI-guided Focal Laser Ablation
Number analyzed (Participants) | 9
Participants | 3

5. Secondary Outcome: Number of Recurrences of Prostate Cancer at the End of 2nd Year Among the Subjects Treated With MRI Guided Focal Laser Interstitial Thermal Ablation
Description: Efficacy is assessed by recurrence rate at end of 2nd year, defined as the number of recurrences divided by the number of patients treated with MRI Guided Focal Laser Interstitial Thermal Ablation
Time Frame: Up to 24 months
Population: Data were not collected/analyzed due to the study termination
Arm/Group | MRI-guided Focal Laser Ablation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | MRI-guided Focal Laser Ablation
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI-guided Focal Laser Ablation (N=9)
Erectile disfunction (Reproductive system and breast disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03634579/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT03634579/ICF_001.pdf